CLINICAL TRIAL: NCT03550066
Title: A Self-Affirmation Intervention to Enhance Patient Outreach for Health System-based Lifestyle Programs for Diabetes Prevention
Brief Title: Patients Engaged in Prevention: Enhancing Outreach to Increase Patient Engagement in Diabetes Prevention
Acronym: PEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CN-14-1871-H; K01DK099404 (NIH); P30DK092924 (NIH)
Record Dates: First submitted 2018-05-14; First posted 2018-06-08 (Actual); Results first posted 2019-08-20 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Preventive Health Services; Health Communication
Keywords: Diabetes, gestational; Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Values affirmation (Experimental): In the values affirmation condition, the health outreach message contained a prompt asking participants to reflect on important personal values.
  Interventions: Behavioral: Values affirmation
- No affirmation (Active Comparator): In the "no affirmation" condition, the health outreach message appeared alone, with no values affirmation.
  Interventions: Behavioral: No affirmation

INTERVENTIONS:
Behavioral: Values affirmation — A health message with a prompt asking participants to reflect on important personal values
  Arms: Values affirmation
Behavioral: No affirmation — A health message alone
  Arms: No affirmation

SUMMARY:
This study examines whether a health message that includes a self-affirmation intervention (where people reflect on values that are important to them) increases acceptance of the message and encourages people to take steps to prevent diabetes, as compared to a health message without the self affirmation intervention.

DETAILED DESCRIPTION:
Background: Despite availability of evidence-based programs for diabetes prevention, few strategies exist to promote patients' interest in them. Strategies should be developed for racial/ethnic minority women with a history of gestational diabetes (GDM), who face exceptionally high risk for chronic diabetes. We previously found that a theory-based outreach message containing a streamlined values affirmation-two sentences prompting individuals to reflect on core personal values-increased women's likelihood of demonstrating interest in a preventive program. Extending this work, this pilot trial tests whether the values affirmation outreach message is as acceptable as (non-inferior to) a standard outreach message among African-American and Latina women.

Methods: Two-arm, parallel-group, randomized trial among English- and Spanish-speaking minority women with prior GDM and overweight/obesity in a healthcare system. Within an online survey, participants are randomized to read an outreach message promoting an existing preventive program. The message contains either a values affirmation (intervention condition) or no affirmation (control condition).

ELIGIBILITY:
Inclusion Criteria:

* History of gestational diabetes
* Body mass index ≥25 kg/m2
* English or Spanish language

Exclusion Criteria:

* Current diabetes
* Current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan D Brown, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northern California, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Values Affirmation | No Affirmation
Started | 49 | 41
Completed | 49 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Affirmation: A health message presented alone, with no values affirmation
- Total: Total of all reporting groups
Arm/Group | Values Affirmation | No Affirmation | Total
Number analyzed (Participants) | 49 | 41 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 41 | 90
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (5.5) | 37.0 (5.2) | 36.5 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 41 | 90
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic Black/African American | 11 | 13 | 24
  Race/Ethnicity: Hispanic/Latina | 36 | 26 | 62
  Race/Ethnicity: More than one race/ethnicity | 2 | 1 | 3
  Race/Ethnicity: Not reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 49 | 41 | 90

OUTCOME MEASURES:

1. Primary Outcome: Acceptance of Health Message
Description: Index of message acceptance: Persuasiveness (rated on a 7-point scale from not at all (1) to very (7), with higher mean scores corresponding to greater persuasiveness)
Time Frame: Up to 2 weeks
Population: Analytic sample, after excluding participants with current diabetes or those already participating in a preventive program
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Values Affirmation | No Affirmation
Number analyzed (Participants) | 45 | 39
units on a scale | 5.5 (0.9) | 5.4 (1.2)
Statistical Analysis 1: Comparison: Values Affirmation vs No Affirmation; Test type: Non-Inferiority — The non-inferiority limit, d, is selected as the largest difference that is clinically acceptable. Here the non-inferiority limit is d=.6 (a medium to large effect size); p = 0.18, t-test, 2 sided — Threshold for statistical significance: <.05

2. Secondary Outcome: Diabetes Prevention Behavior: Information Seeking
Description: Seeking information about prevention
Time Frame: Up to 2 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Values Affirmation | No Affirmation
Number analyzed (Participants) | 45 | 39
Participants | 30 | 30

3. Secondary Outcome: Diabetes Prevention Behavior: Intention
Description: Behavioral intention to engage in, or seeking information about preventive health services
Time Frame: Up to 2 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Values Affirmation | No Affirmation
Number analyzed (Participants) | 45 | 39
Participants | 32 | 34

ADVERSE EVENTS:
Time Frame: 1 month
Description: A priori, few risks were expected, with little to no risk of serious adverse events or mortality. Participants were given contact information to report any concerns about their safety and welfare.
Arm/Group | Values Affirmation | No Affirmation
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/41
Other Adverse Events (participants affected / at risk) | 0/49 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT03550066/Prot_SAP_000.pdf